CLINICAL TRIAL: NCT05629780
Title: Temporal Changes in Plasma Lactate Concentration in Critically Ill Patients With Septic Shock Treated With Restrictive Compared to Standard Fluid Therapy
Brief Title: Temporal Changes of Lactate in CLASSIC Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Collabortation for Research in Intensive Care (CRIC) (Unknown); European Society of Intensive Care Medicine (Other); Region Stockholm (Other Government); The Scandinavian Society of Anaesthesiology and Intensive Care Medicine (SSAI) (Unknown)
Responsible Party: Principal Investigator, Jonathan Grip, Principal Investigator, PhD, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Dnr 2021-06283-02
Record Dates: First submitted 2022-11-14; First posted 2022-11-29 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Intervention Model Description: This is a retrospective analysis of patients recruited to an interventional multicenter trial.
Who Masked: Investigator
Masking Description: All patients are included and analyzed for outcomes in the CLASSIC trial. The allocation and amount of fluids received for the included subjects are blinded for the investigator at the time point of analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative (Experimental): Resuscitation fluids were only given under certain pre-defined criteria
  Interventions: Drug: Resuscitation fluid
- Traditional (liberal) (No Intervention): Patients were treated with standard of care for each site with regards to recuscitation fluids.

INTERVENTIONS:
Drug: Resuscitation fluid — Cristalloid fluids given as a resuscitational intervention
  Arms: Conservative

SUMMARY:
This study aim to examine if randomization to different treatment strategies had any effect on the time to normalization of lactate in intensive care patients treated for septic shock.

DETAILED DESCRIPTION:
This is a retrospective analysis of a subset of patients included in the Conservative versus Liberal Approach to fluid therapy of Septic Shock in Intensive Care (CLASSIC) trial.

In the CLASSIC trial patients with septic shock were randomized to either traditional (liberal) strategy for fluid treatment or a more conservative regimen. The study was an international multicenter clinical trial (clinicaltrials.gov NCT03668236), and results were published in New England Journal of Medicine in June 2022 (DOI: 10.1056/NEJMoa2202707).

In this substudy the investigator extract all lactate values for the study period from all patients included from Karolinska University Hospital, Sundsvall and Södersjukhuset (Sweden), participating centers on Zealand (Denmark), and Plzen University Hospital (Czech Republic). Baseline data, treatment allocation and amount of fluids administered are collected as well as outcome from CLASSIC study.

Primary outcome is time to lactate normalization (< 2mmol/L). Secondary outcome is lactate concentration over the first 72 hours (as peak lactate for the time intervals 0-3, 3-6, 6-12, 12-24 and then each 12h-period between 24 and 72 hours).

The subgroup with blood lactate > 4mmol/L will be analyzed separately for the same end points.

Time to resolution of hyperlactatemia will be modelled with a competing risks regression. Death and discharge will be competing outcomes, and administrative censoring imposed 72 hours after randomisation.

Factors associated with time to lactate normalization will be examined through regression analysis. Factors that show a relationship on univariate analysis will be included in a multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* Participation in CLASSIC trial in any of the participating centres

Exclusion Criteria:

* Lack of sufficient data for analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 777 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
Time to resolution of hyperlactemia | 72 hours
  Blood lactate < 2.0 mmol/L

SECONDARY OUTCOMES:
Temporal changes in lactate concentrations over time | 72 hours
  Difference in blood lactate at during the first 72h from enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meyhoff TS, Hjortrup PB, Wetterslev J, Sivapalan P, Laake JH, Cronhjort M, Jakob SM, Cecconi M, Nalos M, Ostermann M, Malbrain M, Pettila V, Moller MH, Kjaer MN, Lange T, Overgaard-Steensen C, Brand BA, Winther-Olesen M, White JO, Quist L, Westergaard B, Jonsson AB, Hjortso CJS, Meier N, Jensen TS, Engstrom J, Nebrich L, Andersen-Ranberg NC, Jensen JV, Joseph NA, Poulsen LM, Herlov LS, Solling CG, Pedersen SK, Knudsen KK, Straarup TS, Vang ML, Bundgaard H, Rasmussen BS, Aagaard SR, Hildebrandt T, Russell L, Bestle MH, Schonemann-Lund M, Brochner AC, Elvander CF, Hoffmann SKL, Rasmussen ML, Martin YK, Friberg FF, Seter H, Aslam TN, Adnoy S, Seidel P, Strand K, Johnstad B, Joelsson-Alm E, Christensen J, Ahlstedt C, Pfortmueller CA, Siegemund M, Greco M, Radej J, Kriz M, Gould DW, Rowan KM, Mouncey PR, Perner A; CLASSIC Trial Group. Restriction of Intravenous Fluid in ICU Patients with Septic Shock. N Engl J Med. 2022 Jun 30;386(26):2459-2470. doi: 10.1056/NEJMoa2202707. Epub 2022 Jun 17. PMID 35709019

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-12-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT05629780/SAP_000.pdf